CLINICAL TRIAL: NCT01406743
Title: PARAMETRES GLOBAUX DE REFERENCE DU RACHIS CALCULES SUR DES PATIENTS ASYMPTOMATIQUES PAR IMAGERIE EOS™
Brief Title: Spine Reference Parameters on EOS Imaging
Acronym: EOS-SPINE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/26
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers
Keywords: Spine and pelvis parameters; Sagittal balance; Database

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EOS™ Acquisition
  Interventions: Device: EOS™ Acquisition

INTERVENTIONS:
Device: EOS™ Acquisition — Double Incidence Postero Anterior and Lateral full body low-dose X-ray acquisition on EOS™ device following SOP of the service of radiology.

SUMMARY:
The lumbar pain caring consists from a 3D reconstruction of the spine obtained to scan or radiography, determining the lumbar pain cause and gravity, to propose a conservative treatment in first intention or a adapted spine surgery in first or second intention (Fritzell and al ., on 2001).

The analysis and the correction of postural disorders pass inevitably by a good knowledge of the not pathological posture. The validation of the acquisition 2D / 3D reconstruction by EOS ™ technology demonstrated its interest for the diagnosis and the lumbar pain caring.

However, the EOS technology ™ is recent and few data were acquired with this technology for healthy population.

So, this clinical study with EOS ™technology would allow to obtain a precise knowledge of the standing skeleton in position (to an asymptomatic adult population), by displaying the gravity constraints on the joints, and the compensation phenomena in normal situation. This functional information for a given age bracket would allow to propose to the patients with lumbar pain, adapted interventions to the gravity constraints considering the skeleton evolution for age bracket.

DETAILED DESCRIPTION:
The main objective of this study is to describe thoraco-lumbar spine characteristics, obtained by EOS ™technology, in a reference population, not presenting spine pathology. It's a monocentric transverse descriptive study. This study allows creating a database of the spine, pelvis and sagittal balance parameters to asymptomatic subjects according to age brackets.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of more than 18 years old
* Both genders
* Woman under efficient contraception (if not menopause)
* EVA < 2 for the rachis (lumbar vertebra and radiculaire),
* Score ODI ≤ 20 %
* Given informed consent
* Subject with French health system

Exclusion Criteria:

* Pregnant or feeding women
* Subject having a follow-up of the back or a regular back pain,
* Subject presenting lower limbs pathology which can have an echo on the rachis such as a length disparity or a flexum
* Subject with spine and pelvis surgery antecedents.
* Person placed under protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subject without spine pathology
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
the profile spine parameters: apex lumbar position | 1 day
the lordosis lower angle, back type according to the ROUSSOULY | 1 day
the sagittal balance parameters | 1 day
the lordosis upper angle, back type according to the ROUSSOULY | 1 day
the pelvis parameters | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles LE HUEC, PU-PH, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- Spine Unit 2, University Hospital, Bordeaux, France

REFERENCES:
- [Background] Borenstein D. Low back pain: epidemiology, etiology, diagnostic evaluation, and therapy. Curr Opin Rheumatol. 1991 Apr;3(2):207-17. PMID 1829622
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Cats-Baril WL, Frymoyer JW. Identifying patients at risk of becoming disabled because of low-back pain. The Vermont Rehabilitation Engineering Center predictive model. Spine (Phila Pa 1976). 1991 Jun;16(6):605-7. doi: 10.1097/00007632-199106000-00001. PMID 1830688
- [Background] Dubousset J, Charpak G, Dorion I, Skalli W, Lavaste F, Deguise J, Kalifa G, Ferey S. [A new 2D and 3D imaging approach to musculoskeletal physiology and pathology with low-dose radiation and the standing position: the EOS system]. Bull Acad Natl Med. 2005 Feb;189(2):287-97; discussion 297-300. French. PMID 16114859
- [Background] Kalifa G, Charpak Y, Maccia C, Fery-Lemonnier E, Bloch J, Boussard JM, Attal M, Dubousset J, Adamsbaum C. Evaluation of a new low-dose digital x-ray device: first dosimetric and clinical results in children. Pediatr Radiol. 1998 Jul;28(7):557-61. doi: 10.1007/s002470050413. PMID 9662585
- [Background] Fritzell P, Hagg O, Wessberg P, Nordwall A; Swedish Lumbar Spine Study Group. 2001 Volvo Award Winner in Clinical Studies: Lumbar fusion versus nonsurgical treatment for chronic low back pain: a multicenter randomized controlled trial from the Swedish Lumbar Spine Study Group. Spine (Phila Pa 1976). 2001 Dec 1;26(23):2521-32; discussion 2532-4. doi: 10.1097/00007632-200112010-00002. PMID 11725230
- [Background] Geijer H, Verdonck B, Beckman KW, Andersson T, Persliden J. Digital radiography of scoliosis with a scanning method: radiation dose optimization. Eur Radiol. 2003 Mar;13(3):543-51. doi: 10.1007/s00330-002-1476-1. Epub 2002 Jun 14. PMID 12594558
- [Background] Glassman S, Gornet MF, Branch C, Polly D Jr, Peloza J, Schwender JD, Carreon L. MOS short form 36 and Oswestry Disability Index outcomes in lumbar fusion: a multicenter experience. Spine J. 2006 Jan-Feb;6(1):21-6. doi: 10.1016/j.spinee.2005.09.004. PMID 16413443
- [Background] Hansen J, Jurik AG, Fiirgaard B, Egund N. Optimisation of scoliosis examinations in children. Pediatr Radiol. 2003 Nov;33(11):752-65. doi: 10.1007/s00247-003-1015-5. Epub 2003 Sep 5. PMID 12961040
- [Background] Legaye J, Duval-Beaupere G, Hecquet J, Marty C. Pelvic incidence: a fundamental pelvic parameter for three-dimensional regulation of spinal sagittal curves. Eur Spine J. 1998;7(2):99-103. doi: 10.1007/s005860050038. PMID 9629932
- [Background] Pellise F, Hernandez A, Vidal X, Minguell J, Martinez C, Villanueva C. Radiologic assessment of all unfused lumbar segments 7.5 years after instrumented posterior spinal fusion. Spine (Phila Pa 1976). 2007 Mar 1;32(5):574-9. doi: 10.1097/01.brs.0000256875.17765.e6. PMID 17334293
- [Background] Rossignol M, Suissa S, Abenhaim L. Working disability due to occupational back pain: three-year follow-up of 2,300 compensated workers in Quebec. J Occup Med. 1988 Jun;30(6):502-5. PMID 2969044
- [Background] Roussouly P, Berthonnaud E, Dimnet J. [Geometrical and mechanical analysis of lumbar lordosis in an asymptomatic population: proposed classification]. Rev Chir Orthop Reparatrice Appar Mot. 2003 Nov;89(7):632-9. French. PMID 14699309
- [Background] Spengler DM, Bigos SJ, Martin NA, Zeh J, Fisher L, Nachemson A. Back injuries in industry: a retrospective study. I. Overview and cost analysis. Spine (Phila Pa 1976). 1986 Apr;11(3):241-5. doi: 10.1097/00007632-198604000-00010. PMID 2940707
- [Background] Scientific approach to the assessment and management of activity-related spinal disorders. A monograph for clinicians. Report of the Quebec Task Force on Spinal Disorders. Spine (Phila Pa 1976). 1987 Sep;12(7 Suppl):S1-59. No abstract available. PMID 2961086
- [Background] Tournier C, Aunoble S, Le Huec JC, Lemaire JP, Tropiano P, Lafage V, Skalli W. Total disc arthroplasty: consequences for sagittal balance and lumbar spine movement. Eur Spine J. 2007 Mar;16(3):411-21. doi: 10.1007/s00586-006-0208-7. Epub 2006 Sep 8. PMID 16960704